CLINICAL TRIAL: NCT03917303
Title: Control Crohn Safe With Episodic Adalimumab Monotherapy as First Line Treatment Study.
Brief Title: Control Crohn Safe Trial
Acronym: CoCroS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL64005.068.18
Record Dates: First submitted 2019-04-05; First posted 2019-04-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Multicenter randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab (Active Comparator): Episodic adalimumab monotherapy as first line treatment for 6 months
  Interventions: Drug: Adalimumab
- Standard step-up care (Active Comparator): Step-up care as first line treatment, starting with corticosteroids.
  Interventions: Drug: standard step-up care

INTERVENTIONS:
Drug: Adalimumab — episodic treatment with subcutaneous adalimumab for 6 months
  Other Names: Humira
  Arms: Adalimumab
Drug: standard step-up care — conventional step-up care starting with corticosteroids
  Arms: Standard step-up care

SUMMARY:
Crohn's disease (CD) is a chronic disease with a heterogeneous clinical presentation, relapse rate and treatment response. Insufficient control of mucosal inflammation results in irreversible bowel damage and complications and at present no markers are available to predict such a complicated disease course at diagnosis. Therefore, to prevent overtreatment of low risk patients, step-up treatment with subsequent introduction of corticosteroids, thiopurines maintenance and TNF-blockers if a previous category fails is standard care. Combination treatment with thiopurines and a TNF-blocker is more effective than monotherapy but associated with a higher risk for infectious complications. Landmark studies convincingly showed an improved long-term outcome if the TNF-blocker infliximab is introduced early after diagnosis. The standard step-care approach thus prolongs steroid exposure and delays start of disease modifying biologicals in high risks patients. Given the higher efficacy of combination therapy with a thiopurine of infliximab and potential allergic reactions and lower response rates after re-initiation of this chimeric biological, temporary monotherapy with this TNF-blocker has not been studied as first line treatment before. Adalimumab is a humanised monoclonal antibody and subsequently, combination therapy of adalimumab + thiopurines has only a marginal effect on anti-drug anti-body formation. Furthermore, combination therapy with adalimumab does not enhance the clinical response. Therefore, periodic treatment with adalimumab in combination with close monitoring after drug-discontinuation, in newly diagnosed CD might improve outcome, reduce drug-related side effects while still preventing overtreatment.

The aim of this study is to compare the long-term efficacy and safety of periodic adalimumab as initial treatment in newly diagnosed CD patients compared to standard step-care with corticosteroid/budesonide as the initial treatment

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed CD patients or CD patients with a flare, visiting the outpatient clinic or endoscopy ward of the participating centres
* CD diagnosis according to ECCO-guidelines + complete ileo-colonoscopy + complete small bowel imaging at diagnosis (MRI or CT-enterography )
* Naïve to biologicals
* Sufficient knowledge of Dutch language
* 18 years old ≤ 70 years old
* Smartphone with internet access
* Use of myIBDcoach or willingness to start using myIBDcoach

Exclusion Criteria:

* Use of prednisone for longer than 4 weeks in the year before screening
* Use of budesonide (≥6 mg daily) for a duration longer than 3 months in the year before screening
* Use of thiopurines in the 3 years before screening
* Indication for primary treatment with biologicals or surgery
* Malignancy in 5 years before treatment. Exception is adequately treated non-melanoma skin cancer
* Contra-indication for TNF-blockers or immunosuppressive agents
* Contra-indication for MRI- and CT-enterography
* Patients with short bowel syndrome or an ostomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of yearly-quarters of corticosteroid free remission as a measure of treatment efficacy | at week 96
  Remission is defined as combined clinical (MIAH scores (≤3)) and biochemical (C-reactive protein ≤5 mg/L (i.e. within normal range) and fecal calprotectin ≤ 200 μg/g) remission.

SECONDARY OUTCOMES:
Cumulative structural bowel damage as a measure of disease progression | at week 96
  Disease progression on MRI-enterography based on the Lémann score (Crohn's Disease Digestive Damage Score); the Lémann score is an instrument to measure cumulative structural bowel damage in Crohn's disease. The score takes into account the damage location (upper digestive tract, small bowel, colon/rectum and anal/perianal), extent and severity.
  Grades 0 (normal) to 3 (maximal) are given to each segment of the digestive tract, with grade 3 representing the most damage, or resection/bypass.
Incidence of drug related serious adverse events | at week 24, 48 and 96
  Drug related serious adverse events
Incidence of serious disease related adverse events | at week 24, 48 and 96
  Crohn disease related hospitalisation and surgery
Integer amount of direct health care costs (in €) | at week 96
  Direct costs include expenses for medication, diagnostic procedures, number of outpatient clinic visits, hospitalisations and surgeries.
  Direct costs will be combined with indirect costs to report total health care costs.
Integer amount of indirect health care costs (in €) | at week 96
  Indirect costs consist of costs due to presenteeism and absenteeism and are assessed by questionnaires in the telemedicine tool myIBDcoach used for monitoring of IBD patients.
  Indirect costs will be combined with direct costs to report total health care costs.
Corticosteroid use | at week 24, 48 and 96
  Cumulative corticosteroid dose
Endoscopic remission as assessed by SES-CD | at week 24
  Proportion of endoscopic remission based on SES-CD (simple endoscopic score for CD). Endoscopic remission is defined as a score below 3 and the absence of ulcers.
Time to remission | at week 96
  Time to remission
Quality of life as assessed by QoL EQ-5D-5L questionnaire | at week 24, 48 and 96
  Quality of life as assessed by the QoL EQ-5D-5L questionnaire in which the level of severity is chosen for five domains (mobility, self-care, usual activities, pain, anxiety/depression).
  A higher level (maximal 5) indicates more severe problems in that particular domain.

CONTACTS AND LOCATIONS:
Overall Officials: M J Pierik, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (6):
- Netherlands (6):
  - Maastricht University Medical Centre+, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Laurentius Ziekenhuis, Roermond
  - Zuyderland Medical Center, Sittard
  - Máxima Medisch Centrum, Veldhoven
  - VieCuri, Venlo

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers on demand. Patients will be asked to give informed consent to share the collected data with third parties for future research.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Janssen L, Romberg-Camps M, van Bodegraven A, Haans J, Aquarius M, Boekema P, Munnecom T, Brandts L, Joore M, Masclee A, Jonkers D, Pierik M. Control Crohn Safe with episodic adalimumab monotherapy as first-line treatment study (CoCroS): study protocol for a randomised controlled trial. BMJ Open. 2021 May 4;11(5):e042885. doi: 10.1136/bmjopen-2020-042885. PMID 33947729